CLINICAL TRIAL: NCT06479746
Title: Emotional Support Given at Birth to Women Effect on Birth Duration, Perception and Fear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Sukran Ertekin Pinar, Assoc. Prof. Dr., Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TR SİVAS 05
Record Dates: First submitted 2024-06-24; First posted 2024-06-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: First Pregnancy
Keywords: Birth; Emotional support; Birth perception; Fear of birth; Birth duration
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emotional support group (Experimental): Empathetic approach, listening to the feelings and thoughts, welcoming the woman's behavior and expressions, telling her that she is breathing correctly, etc.), not judging the woman, being honest, using a soft and calm tone of voice, taking the baby or asking her opinion, encouraging her to endure the birth process, touching the woman and making physical contact, allowing her to practice her beliefs, showing the baby to the mother as soon as it is born and placing it in her arms.
  Interventions: Behavioral: Emotional support
- Standard of care Group (No Intervention): The control group did not receive any treatment.

INTERVENTIONS:
Behavioral: Emotional support — Emotional support helps the woman giving birth effectively, meets her emotional needs and expectations, ensures her comfort, improves birth outcomes, increases her self-esteem, ensures a positive birth experience and facilitates her transition into the role of motherhood.
  Other Names: Control Group
  Arms: Emotional support group

SUMMARY:
Introduction: Women begin to experience fear long before birth, and the reason for their fear may be related to their baby, themselves, their partner/relatives, and the healthcare professional. Fear can disrupt the natural process of birth, prolong the stages of birth and cause postpartum complications.The research was conducted to determine the effect of emotional support given during birth on the woman's birth duration, perception and fear.

Methods:The population of the randomized controlled experimental study consisted of nulliparous women who applied for normal spontaneous birth to the Birth Unit of a State Hospital in the Central Anatolia Region of Turkey (40 experimental subjects, 40 control subjects).

DETAILED DESCRIPTION:
Introduction: Women begin to experience fear long before birth, and the reason for their fear may be related to their baby, themselves, their partner/relatives, and the healthcare professional. Fear can disrupt the natural process of birth, prolong the stages of birth and cause postpartum complications.Minimizing the fears experienced during birth can lead to more successful and comfortable births, a complication-free birth and less pain for both the woman and the baby.Therefore, emotional support from healthcare professionals is important.

Aim: The research was conducted to determine the effect of emotional support given during birth on the woman's birth duration, perception and fear.

Methods:The population of the randomized controlled experimental study consisted of nulliparous women who applied for normal spontaneous birth to the Birth Unit of a State Hospital in the Central Anatolia Region of Turkey (40 experimental subjects, 40 control subjects).While emotional support practices and standard care were applied to women in the experimental group, only standard care practices were applied to women in the control group. Data were collected using the Personal Information Form, Wijma Birth Expectation/Experience Scale (W-DEQ) Version A, Wijma Birth Expectation/Experience Scale (W-DEQ) Version B, and Women's Perceptions of Supportive Care Provided at Birth Scale.The forms were applied twice to women applying for birth: during labor (first follow-up) and the second follow-up within 2-4 hours after birth. Number and percentage distribution, chi-square test, t test in independent groups, Mann-Whitney U test, Wilcoxon test, and Cohen d test were used in the evaluation of the data.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous,
* Between the ages of 18-35,
* Admitted to the delivery room for normal spontaneous vaginal birth,
* Do not have any physical health problems for themselves or their baby,
* Does not have a diagnosed mental illness,
* Not having a risky pregnancy,
* Able to speak and read Turkish,
* Cervical dilatation of 4 cm or more,
* Women who were willing to participate in the study were included in the study.

Exclusion Criteria:

-Multiparity

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Wijma Delivery Expectancy/Experience Questionnaire version A (W-DEQ-A) | Baseline
  The W-DEQ-A is a validated, to determine the level of birth fear experienced by pregnant women.Answers in the scale are numbered from 0 to 5 and are in a six-point Likert type. The minimum score that can be obtained from the scale is 0, and the maximum score is 165.
Women's Perceptions Scale on Supportive Care Provided at Birth | Baseline
  The scale, which consists of 33 items, has three sub-dimensions: "comforting, informing and disturbing behaviors". Answers in the scale are numbered from 1 to 4 and are in a four-point Likert type. The minimum score that can be obtained from the scale is 33, and the maximum score is 132.

SECONDARY OUTCOMES:
Wijma Birth Expectation/Experience Scale (W-DEQ) Version B | Within 2-4 hours after birth
  W-DEQ-B was developed to evaluate women's fear of birth during their own birth experiences in the postpartum period. Responses on the scale are numbered from 1 to 6 and are in a six-point Likert type. The minimum score that can be obtained from the scale is 33 and the maximum score is 198.
Women's Perceptions Scale on Supportive Care Provided at Birth | Within 2-4 hours after birth
  The scale, which consists of 33 items, has three sub-dimensions: "comforting, informing and disturbing behaviors". Answers in the scale are numbered from 1 to 4 and are in a four-point Likert type. The minimum score that can be obtained from the scale is 33, and the maximum score is 132.

CONTACTS AND LOCATIONS:
Overall Officials: Sukran Ertekin Pinar, Principal Investigator — Cumhuriyet University
Locations (1):
- Sukran Ertekin Pinar, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.